CLINICAL TRIAL: NCT01704599
Title: A Single-Center, Open-Label Study to Assess the Effects of the Addition of Modulators of Homocysteine to Adalimumab Therapy in the Treatment of Moderate to Severe Plaque Psoriasis Evaluated With the PASI, PGA and DLQI
Brief Title: Addition of Modulators of Homocysteine to Adalimumab Therapy in the Treatment of Moderate to Severe Plaque Psoriasis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: side effect and poor clinical outcome
Sponsor: Wayne State University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Peter J. Aronson, MD, Assistant Professor Department of Dermatology, Wayne State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dermatology 1104009591
Record Dates: First submitted 2012-10-03; First posted 2012-10-11 (Estimated); Results first posted 2015-02-04 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-01

CONDITIONS: Psoriasis
Keywords: Psoriasis; Adalimumab; B vitamins; Homocysteine; Folic acid; Cyanocobalamin; Pyridoxine; Vitamin B6; Vitamin B9; Vitamin B12
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab; Vitamin B 6; Pyridoxine; Folic Acid; Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Humira then Humira plus 3 B vitamins (Experimental): Humira then Humira plus 3 B vitamins
  The only arm: After 16 weeks on adalimumab, modulators of homocysteine (oral vitamin B12, oral vitamin B6 or pyridoxine, and oral folic acid) will be added to adalimumab therapy for an additional 12 weeks. At end of this therapy can stop or continue. Telephone call day 70 after formal end of in person study the investigators will assess general health of each subject.
  Interventions: Drug: Humira Then Humira plus 3 B vitamins

INTERVENTIONS:
Drug: Humira Then Humira plus 3 B vitamins — Humira alone for 16 weeks then Humira plus 100 mg daily pyridoxine, 5 mg daily folic acid and 1000 mcg daily cyanocobalamin
  Other Names: Humira; Adalimumab; Vitamin B6; Pyridoxine; Vitamin B9; Folic Acid; Vitamin B12; Cyanocobalamin

SUMMARY:
Vitamins modulating homocysteine affect both TNF-alpha, vascular endothelial growth factor, and theoretically enhance the anti-inflammatory version of NOS thus hopefully increasing the efficacy and reducing the chance of some toxicities of adalimumab as determined by blood testing and EKGs.

DETAILED DESCRIPTION:
This is a pilot study designed to evaluate whether addition of oral vitamin B12, vitamin B6, and folic acid to the use of adalimumab for psoriasis leads to further improvement of a patient's psoriasis and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* adults 18 or older
* moderate to severe plaque psoriasis (>10% BSA)
* Negative pregnancy test within 7 days before first dose of adalimumab in all women (except surgically sterile or 5 years postmenopausal)
* subject must sign/date appropriate written informed consent&HIPAA authorization
* Sexually active subjects of childbearing potential must agree to use medically acceptable contraception during screening and throughout the study
* no evidence of active or latent tuberculosis based on a negative PPD skin test performed at screening, or within one year of starting this study. Patients with documentation of adequately treated TB may be enrolled
* Patients PPD positive and CXR negative can be enrolled if they finish appropriate INH prophylaxis prior to enrollment
* be willing and able to self-administer subcutaneous injections or to have a qualified person available to administer these injections
* agrees to comply with protocol requirements, attend all regularly study visits and is considered to be a good study subject
* meets concomitant medication washout requirements
* willing to use only allowed psoriasis medications and treatments and agree not to start any topical, systemic, or phototherapy for psoriasis during the study period
* adalimumab naïve

Exclusion Criteria:

* erythrodermic, pustular, or guttate psoriasis
* skin conditions other than psoriasis that would interfere with study-related psoriasis evaluations
* known sensitivity to any component of the study medications
* Evidence of active infections such as fevers, chills, sweats, or history of untreated Lyme disease and active severe infections within 4 weeks before screening visit, or between the screening and Week 0 visits
* history of listeriosis, untreated TB, persistent or active infections requiring hospitalization or treatment with IV antibiotics, IV antiretrovirals, or IV antifungals within 30 days of baseline, OR oral antibiotics, antivirals, or antifungals for purpose of treating infection, within 14 days of baseline
* positive PPD and positive chest x-ray for latent or active tuberculosis
* positive PPD and negative chest x-ray that have not completed appropriate INH prophylaxis
* On immune compromising drug or history of immune compromising disorder or immunodeficiency
* poorly controlled medical condition including, not limited to, unstable cardiovascular disease, poorly controlled diabetes, recent stroke, history of recurrent infections, or any condition for which, in the opinion of the investigators, participation in the study would place the subject at risk
* hx. congestive heart failure
* hx. demyelinating CNS disease
* History of malignancy (other than previously treated localized carcinoma in situ of the cervix or previously treated nonmelanoma skin cancer)
* history of or ongoing drug or alcohol abuse
* past or present psychiatric morbidity which may compromise the study
* Pregnant women, nursing mothers, or planning to become pregnant during study or within 150 days after last dose of study medication. Males planning pregnancy with spouse/partner while in study are to be excluded
* plans to receive any live vaccines during study
* history of liver disease
* Current enrollment in another clinical study/treatment with other experimental drug or approved therapy for experimental use within 30 days prior to Week 0
* previous enrollment in this study
* cannot commit to all assessments required by the protocol
* disorder that compromises the subject to give written informed consent and/or comply with study procedures
* considered by the investigators to be unsuitable candidate
* cannot comply with the protocol washout requirements
* on folic acid in doses over than the minimal daily requirements
* on vitamins higher than minimal daily requirements (multivitamins are allowed)
* colon polyps or cancer
* prior adalimumab therapy
* on screening plasma Vascular Endothelial Growth Factor level is 140 pg/ml or more

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-01; Primary Completion 2013-06 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Aronson, MD, Principal Investigator — Department Dermatology Wayne State University

REFERENCES:
- [Background] Aronson PJ, Malick F. Towards rational treatment of severe psoriasis in alcoholics: report of two cases. J Drugs Dermatol. 2010 Apr;9(4):405-8. PMID 20514802
- [Background] Moat SJ, Madhavan A, Taylor SY, Payne N, Allen RH, Stabler SP, Goodfellow J, McDowell IF, Lewis MJ, Lang D. High- but not low-dose folic acid improves endothelial function in coronary artery disease. Eur J Clin Invest. 2006 Dec;36(12):850-9. doi: 10.1111/j.1365-2362.2006.01739.x. PMID 17087779
- [Background] Li W, Zheng T, Wang J, Altura BT, Altura BM. Extracellular magnesium regulates effects of vitamin B6, B12 and folate on homocysteinemia-induced depletion of intracellular free magnesium ions in canine cerebral vascular smooth muscle cells: possible relationship to [Ca2+]i, atherogenesis and stroke. Neurosci Lett. 1999 Oct 22;274(2):83-6. doi: 10.1016/s0304-3940(99)00683-7. PMID 10553943
- [Background] Lewis V, Finlay AY. 10 years experience of the Dermatology Life Quality Index (DLQI). J Investig Dermatol Symp Proc. 2004 Mar;9(2):169-80. doi: 10.1111/j.1087-0024.2004.09113.x. No abstract available. PMID 15083785
- [Background] Gordon KB, Langley RG, Leonardi C, Toth D, Menter MA, Kang S, Heffernan M, Miller B, Hamlin R, Lim L, Zhong J, Hoffman R, Okun MM. Clinical response to adalimumab treatment in patients with moderate to severe psoriasis: double-blind, randomized controlled trial and open-label extension study. J Am Acad Dermatol. 2006 Oct;55(4):598-606. doi: 10.1016/j.jaad.2006.05.027. Epub 2006 Aug 10. PMID 17010738
- [Background] Genovese MC, Mease PJ, Thomson GT, Kivitz AJ, Perdok RJ, Weinberg MA, Medich J, Sasso EH; M02-570 Study Group. Safety and efficacy of adalimumab in treatment of patients with psoriatic arthritis who had failed disease modifying antirheumatic drug therapy. J Rheumatol. 2007 May;34(5):1040-50. Epub 2007 Apr 15. PMID 17444593
- [Background] Pitarch G, Sanchez-Carazo JL, Mahiques L, Perez-Ferriols MA, Fortea JM. Treatment of psoriasis with adalimumab. Clin Exp Dermatol. 2007 Jan;32(1):18-22. doi: 10.1111/j.1365-2230.2006.02288.x. PMID 17305904
- [Background] Leonardi C, Langley RG, Papp K, Tyring SK, Wasel N, Vender R, Unnebrink K, Gupta SR, Valdecantos WC, Bagel J. Adalimumab for treatment of moderate to severe chronic plaque psoriasis of the hands and feet: efficacy and safety results from REACH, a randomized, placebo-controlled, double-blind trial. Arch Dermatol. 2011 Apr;147(4):429-36. doi: 10.1001/archdermatol.2010.384. Epub 2010 Dec 20. PMID 21173304
- [Background] Stuart PE, Nair RP, Ellinghaus E, Ding J, Tejasvi T, Gudjonsson JE, Li Y, Weidinger S, Eberlein B, Gieger C, Wichmann HE, Kunz M, Ike R, Krueger GG, Bowcock AM, Mrowietz U, Lim HW, Voorhees JJ, Abecasis GR, Weichenthal M, Franke A, Rahman P, Gladman DD, Elder JT. Genome-wide association analysis identifies three psoriasis susceptibility loci. Nat Genet. 2010 Nov;42(11):1000-4. doi: 10.1038/ng.693. Epub 2010 Oct 17. PMID 20953189
- [Background] Institute of Medicine (US) Standing Committee on the Scientific Evaluation of Dietary Reference Intakes and its Panel on Folate, Other B Vitamins, and Choline. Dietary Reference Intakes for Thiamin, Riboflavin, Niacin, Vitamin B6, Folate, Vitamin B12, Pantothenic Acid, Biotin, and Choline. Washington (DC): National Academies Press (US); 1998. Available from http://www.ncbi.nlm.nih.gov/books/NBK114310/ PMID 23193625
- [Background] Suarez-Farinas M, Fuentes-Duculan J, Lowes MA, Krueger JG. Resolved psoriasis lesions retain expression of a subset of disease-related genes. J Invest Dermatol. 2011 Feb;131(2):391-400. doi: 10.1038/jid.2010.280. Epub 2010 Sep 23. PMID 20861854
- See also: Search for Humira — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm?fuseaction=Search.DrugDetails
- See also: hypermagnesemia — http://www.emedicine.com/med/topic3383.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were recruited at one of the Two Wayne State University Physician Group Dermatology clinics . Recruitment began Oct 2010 and lasted until 2012
Pre-assignment Details: There were 11 potential subjects analyzed of which 3 were not enrolled prior to study assignment. The 3 did not meet study criteria.
Groups:
- Humira Then Humira Plus 3 B Vitamins: Humira then Humira plus 3 B vitamins
  The one arm: After 16 weeks on adalimumab, modulators of homocysteine (oral vitamin B12, oral vitamin B6 or pyridoxine, and oral folic acid) will be added to adalimumab therapy for an additional 12 weeks. At end of this, therapy can stop or continue . Telephone call day 70 after formal end of in person study the investigators will assess general health of each subject.
  Humira Then Humira plus 3 B vitamins: Humira alone for 16 weeks then Humira plus 100 mg daily pyridoxine, 5 mg daily folic acid and 1000 mcg daily cyanocobalamin
Period: Overall Study
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Started | 8 (Study was started January 22, 2010)
Completed | 7 (11 screened 8 entered study 1 terminated.)
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: 5 male 3 female Adults over age 18 < or = 65 7 Adults over age 65 1
Groups:
- Humira Then Humira Plus 3 B Vitamins: Humira then Humira plus 3 B vitamins
  The only arm: After 16 weeks on adalimumab, modulators of homocysteine (oral vitamin B12, oral vitamin B6 or pyridoxine, and oral folic acid) will be added to adalimumab therapy for an additional 12 weeks. At end of this therapy can stop or continue . Telephone call day 70 after formal end of in person study the investigators will assess general health of each subject.
  Humira Then Humira plus 3 B vitamins: Humira alone for 16 weeks then Humira plus 100 mg daily pyridoxine, 5 mg daily folic acid and 1000 mcg daily cyanocobalamin
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants] — Eleven subjects went for screening: 8 were labelled 'White' though one had an Asian name(From India) and 3 were African American.
  Three subjects failed screening: two Caucasian: one white, one was the 'white' person with the Asian name and one African American.
  Of the 8 who were enrolled, 2 were African American and 6 were Caucasian (white).
  The one enrolled subject who develeoped an SAE before entering the vitamin plus adalimumab part of the study was white.
  The seven who completed the study: 5 Caucasians and 2 African Americans.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 2
    White | 6
    More than one race | 0
    Unknown or Not Reported | 0
number enrolled participants [Number; unit: participants 8] | 8
Adult patients with plaque psoriasis >10% BSA [Number; unit: participants]
  Male | 5
  Female | 3

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With a Categorical Change in Static Physician Global Assessment (sPGA):
Description: Number of participants with a category change in Physician static Global Assessment (sPGA): 7 point score from 0 (clear) to 6 measuring amount of surface covered and plaque qualities: thickness & erythema plus scaling. Dynamic score compares baseline with either improvement/ worsening of the same factors measured in the sPGA using the 0-6 scoring range but focused on change. sPGA at weeks 16 AND 28. dynamic PGA to be categoically measured at.weeks16 and 28.
Time Frame: Week 16 and Week 28
Population: 8 adult participants with moderate to severe plaque psoriasis. 7 had static PGA scores weeks 16 and 28 and one had sPGA but SAE prior to week 16.
Measure: Number; unit: participants
Groups:
- Humira Then Humira Plus 3 B Vitamins: Adults ages 18-65 with moderate to severe plaque psoriasis measured at week 16 after 16 weeks of adalimumab and week 28 after 16 weeks of adalimumab then 12 weeks of adalimumab plus 5 mg folic acid, 100 mg vitamin B6 and 1000 mcg of B12.
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Number analyzed (Participants) | 7
participants
  Improved | 3
  Unchanged | 1
  Worsened | 3

2. Secondary Outcome: Number of Participants With a Categorical DLQI (Dermatology Life Quality Index) Change
Description: DLQI is 10 questions examining impact of skin disease on quality of life: (1) symptoms & feelings (2) daily activities (3) leisure (4) work & school (5) personal relationship (6) treatment. To be administered to adults over 18 years with moderate to severe plaque psoriasis at week 0 (no systemic psoriasis medication);. weeks 16 ( after 16 weeks of adalimumab) and week 28 (after 16 weeks adalimumab then 12 weeks of adalimumab plus daily 5 mg folic acid, 100 mg vitamin B6 and 1000 mcg B12).
Time Frame: Week 16 and Week 28
Population: 8 adults with moderate to severe plaque psoriasis measured at weeks 16 and 28. Seven were measured weeks 16 and 28. One had SAE prior to week 16.
Measure: Number; unit: participants
Groups:
- Humira Then Humira Plus 3 B Vitamins: Adults ages 18-65 years with moderate to severe plaque psoriasis evaluated at week 0 on no systemic psoriasis medication; weeks 16 after 16 weeks adalimumab and 28 after 16 weeks adalimumab then 12 weeks adalimumab plus 5 mg folic acid, 100 mg vitamin B6 and 1000 mcg B12.
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Number analyzed (Participants) | 7
participants
  Improved | 3
  Unchanged | 3
  Worsened | 1

3. Other Pre Specified Outcome: Number of Participants in the Categories of Having and Not Having an Adverse Event
Description: Worsening psoriasis or development or worsening of measured condition or new pathology not seen by week 16 but developed at weeks 28 or first discoved by telephone call day 70 post study:
  AE Humira only
Time Frame: After Week 16 of study
Population: 8 adult participants ages 18-65 with moderate to severe plaque psoriasis. Seven assessed after week 16 and at Week 28 of study and assessed at day 70 post week 28 visit ( the latter by telephone). One subject had SAE prior to vitamin addition.
Measure: Number; unit: participants
Groups:
- Humira Then Humira Plus 3 B Vitamins: Adults ages 18-65 with moderate to severe plaque psoriasis evaluated at after week 16 of study on or after of adalimumab then 12 weeks of adalimumab plus daily 5 mg folic acid, 100 mg vitamin B6 and vitamin B12 or during the 10 weeks after that.
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Number analyzed (Participants) | 7
participants
  No Adverse Event after Week 16 | 2
  Adverse Event Weeks 16-28 | 4
  Adverse event by Day 70 call after Week 28 | 1

4. Other Pre Specified Outcome: Number of Participants in the Categories of Having and of Not Having a Serious Adverse Event (SAE)
Description: A serious adverse event is hosptalization or death or pathology leading to early termination of a participant from the study. This was to be reported at anytime during the 28 week study of adult patients ages 18-65 with moderate to severe plaque psoriasis though categorized by Week 16 (on adalimumab alone, by Week 28 (on adalimuamb plus 3 B vitaminsand by day 70 post Week 28.
Time Frame: By Week 16, by Week 28 and by Day 70 post Week 28.
Population: Adults ages 18-65 with moderate to severe plaque psoriasis.
Measure: Number; unit: participants
Groups:
- Humira Then Humira Plus 3 B Vitamins: Adult 18-65 year old adults with moderate to severe plaque psoriasis with adverse event documented sometime during the 28 week study plus telephone call day 70 post week 28 visit either with knowledge of serious event of adverse event documented from data taken weeks 4 and 16 on adalimumab alone and week 28 after 16 weeks on adalimumab plus 12 weeks on adalimumab and daily 5 mg folic acid, 100 mg vitamin B6 and 1000 mcg B12 and a telephone call day 70 post week 28 study visit and a telephone call day 70 post week 28 visit.
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Number analyzed (Participants) | 8
participants
  No SAE | 7
  SAE by Week 16 | 1
  SAE by Week 28 | 0
  SAE by Day 70 afterWeek 28 | 0

5. Other Pre Specified Outcome: Number of Participants in the Categories of Normalizing, Unchanging and Newly Abnormal Electrocardiograms (EKGs)
Description: An electrocardiogram (EKG) is used to evaluate the electrical activity of the heart by converting this activity into line tracings on paper.. Electrodes (small, plastic patches) are placed at certain locations on the chest, arms, and legs. When the electrodes are connected to an EKG machine by lead wires, the electrical activity of the heart is measured, interpreted, and printed out for the doctor's information and further interpretation. This test was to be administered to adults age 18 or older with moderate to severe plaque psoriasis patients at week 0, 16 and week 28 of this study.
Time Frame: Week 16 and then Week 28 after another 12 weeks on Humira plus vitamins and if early termination
Population: 8 adults with moderate to severe plaque psoriasis. Seven evaluated at weeks 0,16 and 28 for no change in electrocardiogram (EKG) , worsening arrhymia or improvement of arrhythmia at weeks 16 and 28. Five of 8 studied weeks 0,16 and 28; 1 at week 16 and 28. Two (one with the SAE prior to Week 16) did not have EKGs both at weeks 16 and 28.
Measure: Number; unit: participants
Groups:
- Humira Then Humira Plus 3 B Vitamins: Adults ages 18-65 years with moderate to severe plaque psoriasis measured at week 0 on no systemic psoriasis medication; week 16 on adalimumab for 16 weeks and then week 28 after 16 weeks of adalimumab then 12 weeks of adalimumab plus 5 mg folic acid, 100 mg vitamin B6 and 1000 mcg of B12.
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Number analyzed (Participants) | 6
participants
  Normalizing | 1
  Unchanged | 4
  Newly abnormal | 1

6. Secondary Outcome: Number of Participants With Category Change in Serum VEGF (Vascular Endothelial Growth Factorl)
Description: Adult particpants ages 18 or older with moderate to severe plaque psoriasis were to have serum VEGF measured at week 0 on no systemic psoriasis medication then at both weeks 16 on adalimumab and at week 28 on adalimumab plus folic acid, B6 and Vitamin B12. Subjects raniked by BMI week 0 low to high
Time Frame: At Screening visit, Week 16 on Humira, after another 12 weeks on Humira plus vitamins and if early termination
Population: 8 adult subjects age 18-65 with moderate to sefver plaque psoriasis. Five subjects had VEGF levels taken weeks 16 and 28. Three ( one wiht SAE prior to week 16) did not.
Measure: Number; unit: participants
Groups:
- Humira Then Humira Plus 3 B Vitamins: Adults ages 18-65 with moderate to severe plaque psoriasis with subject serum levels to be measured weeks 16 after 16 weeks of adalimumab and week 28 after 16 weeks of adalimumab and then 12 weeks of adalimumab plus daily 5 mg folic acid, 100 mg vitamin B6 and 1000 mcg of vitamin B12.
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Number analyzed (Participants) | 5
participants
  Increased | 4
  Unchanged | 0
  Decreased | 1

7. Other Pre Specified Outcome: Number of Participants in Categories or Increasing and Decreasing Changes Within the CBC (Complete Blood Count)
Description: Change in CBC parameter: white blood count or hemoglobin or hematocrit ( as measured week 16 on adalimumab and at week 28 after 12 more weeks on adalimuamb , folic acid, B6 and B12) in adults ages 18-65 with moderate to severe plaque psoriasis.
Time Frame: Week 16 and Week 28
Population: 8 adult participants with moderate to severe plaque psoriasis. Five had CBCs at both week 16 and week 28. three did not ( one of the 3 had a SAE pripor to week 16)
Measure: Number; unit: participants
Groups:
- Humira Then Humira Plus 3 B Vitamins: Adult subjects ages 18-65 with moderate to severe plaque psoriasis measured at week 0 on no systemic psoriasis medication ,week 16 after 16 wqeeks of adalimumab and week 28 after 16 weeks of adalimumab then 12 weeks of adalimumab plus folic acid 5 mg. vitamin B6 100 mg and vitamin B12 1000 mcg daily assessing CBC with diferential for increase, decrease and no change.
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Number analyzed (Participants) | 5
participants
  WBC increased | 3
  WBC unchanged | 0
  WBC decreased | 2
  Hemoglobin/Hematocrit increased | 3
  Hemoglobin/Hematocrit unchanged | 0
  Hemoglobin/Hematocrit decreased | 2

8. Other Pre Specified Outcome: Number of Participants Within the Categories of Increasing and Decreasing Serum Magnesium
Description: Serum magnesium (Mg) was to be measured at baseline, Week 16 (on adalimumab) and at week 28 (on adalimumab plus folic acid, vitamins B6 and B12) in adult participants age 18 or older with moderate to severe plaque psoriasis.
Time Frame: Weeks 16 and 28
Population: 8 Adults age 18-65 with moderate to severe plaque psoriasis.Five had results both weeks 16 and 28. Three did npot (of these 1 had SAE prior to week 16)
Measure: Number; unit: participants
Groups:
- Humira Then Humira Plus 3 B Vitamins: 8 adult 18-65 year old moderate to severe plaque psoriasis patients with levels measured weeks 0,16 and 28 in 4 subjects; weeks 0 and 16 in one subject, weeks 16 and 28 in one subject and week 0 only in 2 subjects.
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Number analyzed (Participants) | 5
participants
  Increased | 1
  Unchanged | 2
  Decreased | 2

9. Other Pre Specified Outcome: Number of Participants Within the Categories of Increasing and Decreasing Serum Phosphorus
Description: Serum phosphorus (P) levels were to be measured weeks16 and 28 in adult participants age 18 and older with moderate to severe plaque psoriasis at week 0 on no systemic psoriasis medication; week 16 after 16 weeks of adalimumab and at week 28 after 16 weeks of adalimumab plus 12 weeks of adalimumab plus 5 mg folic acid, 100 mg vitamin B6 and 1000 mcg of B12.
Time Frame: Week 16 then Week 28
Population: 8 adults 18-65 years having moderate to severe plaque psoriasis. Five had levels measured at week 16 and and again at week 28 . Three did not . Of the 3 1 had SAE prior to week 16.
Measure: Number; unit: participants
Groups:
- Humira Then Humira Plus 3 B Vitamins: Adults 18-65 all with moderate to severe plaque psoriasis. Week 0 (on no systemic psoriasis medication), Week 16 ( 16 weeks adalimumab), Week 28 ( 16 weeks on adalimumab plus 12 weeks on adalimumab plus 5 mg folic acid, 100 mg B6 and 1000 mcg B12 daily.
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Number analyzed (Participants) | 5
participants
  Increased | 3
  Unchanged | 0
  Decreased | 2

10. Secondary Outcome: Number of Participants Within the Categories of Increasing and Decreasing Serum Homocysteine
Description: Serum homocysteine measured at week 16 after 16 weeks of adalimumab and week 28 after 16 weeks of adalimumaband then 12 weeks of adalimumab plus 5 mg folic acid, 100mg B6 and 1000 mcg of B12 in adults ages 18-65 with moderate to sever plaque psoriasis..
Time Frame: Week 16 and Week 28
Population: 8 adults 18-65 with moderate to severe plaque psoriasis. 4 had levels measured at Week 16 and again at Week 28. Of the 4 not meausres 1 had a SAE prior to Week16.
Measure: Number; unit: participants
Groups:
- Humira Plus 3 B Vitamins: adults 18-65 with plaque psoriasis (moderate to severe) measured at week 0 on no systemic psoriasis medication; week 16 after 16 weeks adalimumab and at 28 weeks after 16 weeks adalimumab plus 12 weeks folic acid, vitamin B6 and B12.
Arm/Group | Humira Plus 3 B Vitamins
Number analyzed (Participants) | 4
participants
  Increased | 1
  Unchanged | 0
  Decreased | 3

11. Secondary Outcome: Number of Participants With Category Change in Vitamin B12 Blood Level
Description: Adult participants 18 years or older with moderate to severe plaque psoriasis were to have serum B12 levels measures Weeks 0 (on no systemic psoriasis medication), 16 (on adalimumab) and week 28 (on adalimumab plus daily 5 mg folic acid, 100 mg vitamin B6 and 1000 mcg B12.
Time Frame: At Week 16 and Week 28
Population: 8 adult participants ages 18-65 with moderate to severe plaque psoriasis. Five of 8 had B12 measured at weeks 16 and 28. Three did not. One of the 3 had SAE prior to week 16.
Measure: Number; unit: participants
Groups:
- Humira Then Humira Plus 3 B Vitamins: Adults ages 18-65 with moderate to severe plaque psoriasis.
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Number analyzed (Participants) | 5
participants
  Increased | 5
  Unchanged | 0
  Worsened | 0

12. Secondary Outcome: Number of Participants Within the Categories of Increasing and Decreasing Serum Vitamin B6 Level
Description: Serum vitamin B6 levels were to be measured weeks16 after 16 weeks adalimumab and at week 28 after 16 weeks adalimumab and 12 weeks on adalimuamb, folic acid 5 mg, b6 100 mg and B12 1000 mcg in adult participants with moderate to sever plque psoriasis.
Time Frame: At Week 16 and Week 28
Population: 8 adults 18-65 with moderate to severe plaque psoriasis measured at weeks 16 and 28. .Four of 8 had levels drawn at weeks 16 and 28. Four did not. Of the four whoi did not one had a SAE prior to Week 16.
Measure: Number; unit: participants
Groups:
- Humira Then Humira Plus 3 B Vitamins: Adults 18-65 years with moderate to severe plaque psoriasis measured at week 16 after 16 weeks adalimumab and week 28 after 28 weeks adalimumab annd 12 weeks on adalimumab, folic acid 5 mg, 100 mg B6 and 1000 mcg B12.
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Number analyzed (Participants) | 4
participants
  Increased | 4
  Unchanged | 0
  Decreased | 0

13. Secondary Outcome: Number of Participants With Category Change in Serum Folic Acid Level.
Description: Serum folic acid level in adults ages 18 and older with mild to moderate plaque psoriasis measured at week 16 after 16 weeks adalimumab and at week 28 after 16 weeks adalimumab plus 12 weeks of adalimumab and daily 5 mg folic acid, 100 mg vitamin B6 and 1000 mcg B12.
Time Frame: Weeks 16 and 28
Population: 8 particpantts with psoriasis. Five had folic acid levels drawn weeks 16 and 28. Three did not (one of the 3 had a SAE prior to week 16).
Measure: Number; unit: participants
Groups:
- Humira Then Humira Plus 3 B Vitamins: Adults ages 18-65 with moderate to severe plaque psoriasis measured at 16 after 16 weeks of adalimumab and week 28 after 16 weeks of adalimumab then 12 weeks of adalimumab and daily 5 mg folic acid 100 mg vitamin B6 and 1000 mcg B12.
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Number analyzed (Participants) | 5
participants
  Increased | 3
  Unchanged | 0
  Decreased | 0
  Not evaluable (if >20 ng/ml only stated as such) | 2

14. Other Pre Specified Outcome: Number of Participants Within the Categories of Elevated and Normal Helicobacter Pylori Antibody
Description: Adult participants age 18 years or older with moderate to severe plaque psoriasis with serum IgG antibodies against Helicobacter pylori bacteria using commercial ELISA assay during the 28 week study.
Time Frame: Week 28 after 16 weeks of Adalimumab then 12 of Adalimumab-Vitamins
Population: 8 adult participants with moderate to severe plaque psoriasis with H. pylori titers measured during the 28 week study.
Measure: Number; unit: participants
Groups:
- Humira Then Humira Plus 3 B Vitamins: 8 adults ages18-65 with moderate to severe plaque psoriasis tested at week 0 on no systemic psoriasis therapy; week 16 after 16 weeks of adalimumab and week 28 after 16 weeks adalimumab plus 5 mg folic acid, 100 mg B6 and 1000 mcg B12.
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Number analyzed (Participants) | 8
participants
  Elevated | 2
  Normal | 6

15. Other Pre Specified Outcome: Number of Participants Within the Categories of Positive Urine Pregnancy Test (Urine Hcg)
Description: Women of childbearing years over age 18 with moderate to severe plaque psoriasis on no systemic therapy at week 0 of study.
Time Frame: At screening
Population: Only 1 of the 8 subjects was a woman of childbearing years during the study.
Measure: Number; unit: participant
Groups:
- Humira Then Humira Plus 3 B Vitamins: One adult psoriasis subject age 23 with moderate to severe plaque psoriasis with pregnanacy test on enrollment on no systemic psoriasis therapy.
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Number analyzed (Participants) | 1
participant
  Negative | 1
  Positive | 0

16. Other Pre Specified Outcome: Number of Participants Within the Categories of Increasing and Decreasing Blood Pressure and Pulse Measures:
Description: Blood pressure is the force the heart exerts against the walls of arteries as it pumps the blood out to the body. The unit of measurement is millimeters of mercury (mm Hg). Pulse is the number of times your heart beats per minute. The unit of measurement is beats per minute (BPM). These test measurements compared in adults with moderate to severe plaque psoriasis week 16 after 16 weeks adalimumab and week 28 after 16 weeks adalimumab plus 5 mg folic acid, 100 mg vitamin B6 and 1000 mcg vitamin B12.
Time Frame: Week 16 and Week 28
Population: of 8 adults with moderate to severe plaque psoriasis, Seven participants were measured at week 16 after 16 weeks adalimumab and at week 28 after 16 weeks adalimumab then 12 weeks of adalimumab plus 5 mg folic acid, 100 mg vitamin B6 and 1000 mcg B12. One who had SAE prior to Week 16 did not..
Measure: Number; unit: participants
Groups:
- Humira Then Humira Plus 3 B Vitamins: Subjects were adults with moderate to severe plaque psoriasis with test to be measured week 0 on no systemic psoriasis medication, week 16 after 16 weeks adalimumab and week 28 after 16 weeks adalimumab plus 5 mg folic acid, 100 mg vitamin B6 and 1000 mcg of vitamin B12.
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Number analyzed (Participants) | 7
participants
  Systolic BP increased | 4
  Systolic BP unchanged | 0
  Systolic BP decreased | 3
  Diastolic BP increased | 5
  Diastolic BP unchanged | 0
  Diastolic BP decreased | 2
  Pulse increased | 5
  Pulse unchanged | 0
  Pulse decreased | 2

17. Other Pre Specified Outcome: Number of Participants Within Categories of Body Temperature Change
Description: Using a thermometer for body temperature on degrees Fahrenheit. Participants to be measured were adults 18 years or older with moderate to severe plaque psoriasis with temperature to be measured at week 16 16 weeks of adalimumab and week 28 after 16 weeks of adalimumab then 12 weeks of adalimumab plus 5 mg folic acid, 100 mg vitamin B6 and 1000 mcg of B12.
Time Frame: Weeks 16 and 28
Population: 8 Subjects. Five had temperatures measured weeks 16 and 28. Three did not (one of the 3 had SAE prior to week16)
Measure: Number; unit: participants
Groups:
- Humira Then Humira Plus 3 B Vitamins: Temperature measurements in adults ages 18-65 with moderate to severe plaque psoriasis at week16 on adalimuamb and week 28 temperatures on adalimumab and daily 5 mg folic acid, 100 mg vitamin B6 and 1000 mcg B12.
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Number analyzed (Participants) | 5
participants
  increased | 2
  unchanged | 2
  decreased | 1

18. Other Pre Specified Outcome: Number of Participants Who Fulfilled the Category of Having Height Measured
Description: Height is the distance from the bottom (soles of feet ) to the top (top of head) of a person when that person is standing in this study using ruler in inches.Participants measured were adults age 18 or older with moderate to severe plaque psoriasis.
Time Frame: Week 0 at Start of Adalimumab
Population: 8 Adults with mild to moderate plaque psoriasis had their height measured at week 0 in inches.
Measure: Number; unit: participants
Groups:
- Humira Then Humira Plus 3 B Vitamins: 8 adults age 18-65 yearswith moderate to severe plaque psoriasis measured at week 0 of study on no systemic psoriasis medication.
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Number analyzed (Participants) | 8
participants
  Measured | 8
  Not measured | 0

19. Other Pre Specified Outcome: Number of Participants Within the Categories of Increasign and Decreasing Body Weight
Description: Weight is how heavy a participant is. Weight in pounds of each study adult participant age 18-65 years with moderate to severe plaque psoriasis measured at weeks 16 and compared to week 28 of study.
Time Frame: Week 16 and Week 28
Population: 8 adults ages 18-65 with moderate to severe plaque psoriasis. Seven of 8 had weights taken weeks 0,4,16 and 28 allowing week16 and 28 analysis. One had weight taken only at weeks 0 and 4.
Measure: Number; unit: participants
Groups:
- Humira Then Humira Plus 3 B Vitamins: Adults ages 18-65 years with moderate to severe plaque psoriasis. Weight measurement were in pounds measured at Weeks 16 and 28.
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Number analyzed (Participants) | 7
participants
  Increased | 2
  Unchanged | 0
  Decreased | 5

20. Primary Outcome: Number of Particpants With a Categorical PASI (Psoriasis Area and Severity Index) Change
Description: PASI: formula based on body surface areas on head/neck, trunk, both arms & legs with disease quality grading induration, scale and erythema on participants ages 18-65 with moderate to severe plaque psoriasis measured at weeks 16 and 28.
Time Frame: Weeks 16 and 28
Population: 8 adults ages 18-65 with moderate to severe plaque psoriasis. Seven of 8 had PASI measured at weeks 16 and 28. One had SAE prior to week 16.
Measure: Number; unit: participants
Groups:
- Humira Then Humira Plus 3 B Vitamins: 8 adults ages 18-65 with moderate to severe plaque psoriasis with PASI measured week 0 on no systemic psoriasis medication, weeks 4 and 16 after 4 and 16 weeks of adalimumab and week 28 after 16 weeks of adalimumab plus 12 weeks of adalimumab and 5 mg folic acid, 100 mg vitamin B6 and 1000 mcg of B12 ranked by calculated Body Mass Index (BMI) week 0.
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Number analyzed (Participants) | 7
participants
  Improved | 4
  Unchanged | 1
  Worsened | 2

21. Post Hoc Outcome: PASI Change Related to Baseline Body Mass Index Above, Below and Equal to 27.3
Description: Change in PASI from Week 16 on adalimumab to Week 28 on adalimumab, folic acid, vitamin B6 and B12 in adults ages 18-65 with moderate to severe plaque psoriasis.
Time Frame: Week 16 and Week 28
Population: 8 Adult subjects ages 18-65 with moderate to severe plaque psoriasis. 7 had PASI data both Week 16 and Week 28. The 1 who did not had SAE prior to Week 16.
Measure: Number; unit: participants
Groups:
- Humira Then Humira Plus 3 B Vitamins: Humira then Humira plus 3 B vitamins
  The only arm: After 16 weeks on adalimumab, modulators of homocysteine (oral vitamin B12, oral vitamin B6 or pyridoxine, and oral folic acid) will be added to adalimumab therapy for an additional 12 weeks. At end of this therapy can stop or continue. Telephone call day 70 after formal end of in person study the investigators will assess general health of each subject.
  Humira Then Humira plus 3 B vitamins: Humira alone for 16 weeks then Humira plus 100 mg daily pyridoxine, 5 mg daily folic acid and 1000 mcg daily cyanocobalamin
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Number analyzed (Participants) | 7
participants
  BMI >27.3 who improved | 4
  BMI >27.3 who worsened | 0
  BMI of 27.3 who were unchanged | 0
  BMI<27.3 who improved | 0
  BMI<27.3 who worsened | 2

22. Post Hoc Outcome: PASI Change in Participants With Baseline VEGF Above 140 pg/ml and in Participants With Normal Baseline VEGF
Description: Baseline VEGF level at week zero related to PASI change Week 16 on adalimumab compared to Week 28 after additonal 12 weeks of adalimumab plus folic acid, vitamin B6 and B12 in adult psoriasis patients ages 18-65 with moderate to severe plaque psoriasis.High levels were greater than or equal to 140 pg/ml. Normal VEGF was below this level.
Time Frame: Week 16 and Week 28
Population: 8 adult participants with moderate to severe plaque psoriasis ages 18 to 65. Seven were analyzed. The one not analyzed had SAE prior to week16.
Measure: Number; unit: participants
Groups:
- Humira Then Humira Plus 3 B Vitamins: Humira then Humira plus 3 B vitamins
  The one arm: After 16 weeks on adalimumab, modulators of homocysteine (oral vitamin B12, oral vitamin B6 or pyridoxine, and oral folic acid) will be added to adalimumab therapy for an additional 12 weeks.
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Number analyzed (Participants) | 7
participants
  PASI improved with high VEGF | 1
  PASI Worsened with high VEGF | 2
  PASI Unchanged with normal VEGF | 1
  PASI Improved with normal VEGF | 3
  PASI Worsened with normal VEGF | 0

23. Post Hoc Outcome: Psoriasis Change in Participants With High H. Pylori Titers and With Normal Titers.
Description: Change in PASI from Week 16 after 16 weeks of adalimumab to Week 28 after another 12 weeks of adalimumab plus folic acid, vitamins B6 and B12 and Change reported by telephone 70 days after week 28
Time Frame: Week 16 to Week 28 and Week 28 to post study day 70
Population: 8 Adults ages 18-65 with moderate tosevere plaque psoriasis. 7 subjects studied. The 8th had SAE prior to Week 16.
Measure: Number; unit: participants
Groups:
- Humira Then Humira Plus 3 B Vitamins: Humira then Humira plus 3 B vitamins
  The one arm: After 16 weeks on adalimumab, modulators of homocysteine (oral vitamin B12, oral vitamin B6 or pyridoxine, and oral folic acid) will be added to adalimumab therapy for an additional 12 weeks. At end of this, therapy can stop or continue . Telephone call day 70 after formal end of in person study the investigators will assess general health of each subject.
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Number analyzed (Participants) | 7
participants
  high titer worsened | 1
  high titer improved then worsened day 70 | 1
  normal titer improved | 3
  normal titer unchanged then improved day 70 | 1
  normal titer worsened | 1

24. Post Hoc Outcome: EKG Categoryy Changes Related to Homocysteine Changes
Description: Change in EKG ( normalize, unchanged, became abnormal) when homocysteine (Hcy) increased or decreased from week 16 on adalimumab to week 28 on adalimumab plus folic acid, vitamins B6 and B12 in adault psoriasis patients ages 18-65 with moderate to severe plaque psoriasis.
Time Frame: Week 16 to Week 28
Population: 8 adults with moderate to severe plaque psoriasis ages 18-65. 4 were studied. Four were not because homocysteine levels at both Week16 nd 28 were not drawn(1 of the 4 had SAE prior to Week 16).
Measure: Number; unit: participants
Groups:
- Humira Then Humira Plus 3 B Vitamins: Humira then Humira plus 3 B vitamins
  The one arm: After 16 weeks on adalimumab, modulators of homocysteine (oral vitamin B12, oral vitamin B6 or pyridoxine, and oral folic acid) will be added to adalimumab therapy for an additional 12 weeks (week 28).
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Number analyzed (Participants) | 4
participants
  normalize when Hcy increased | 1
  unchanged when Hcy decreased | 2
  became abnormal when Hcy decreased | 1

ADVERSE EVENTS:
Time Frame: 2010-2013
Description: On Humira alone: WBC elevation, Non specific st-t wave change and Left axis deviation. .
Groups:
- Humira Then Humira Plus 3 B Vitamins: Pneumonia while on adaimumab and before the adalimumab plus B vitamins were begun.prior to vitamins
Arm/Group | Humira Then Humira Plus 3 B Vitamins
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 3/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Humira Then Humira Plus 3 B Vitamins (N=8)
Pneumonia (Infections and infestations) | 1 (1) — Pneumonia while on adalimumab before vitamins.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Humira Then Humira Plus 3 B Vitamins (N=7)
left axis deviation (Cardiac disorders) | 2 (2) — EKG change one on Humira alone the otehr on drug plus vitamines (note: the fisrt subject with left axis deviation became normal after on vitamins were added)
psoriasis flare (Skin and subcutaneous tissue disorders) | 3 (3) — 2 subjects' psoriasis worsened by PASI after vitamins added to adalimumab (1 one also by BSA and one also by DLQI) one additional flare noted post study day 70 still on adalimumab.
Elevated White blood count (Blood and lymphatic system disorders) | 1 (1) — Occurred while on Humira alone in 1 subject.
elevated Helicobacter pyori antibody (Infections and infestations) | 1 (1) — New elevation after week 0 in 1 subject after vitamins added to Humira
nonspecific st-t wave changes (Cardiac disorders) | 1 (1) — Occurred in 1 subject on Humira alone.

LIMITATIONS AND CAVEATS:
Early termination due to high amount of combination of side effects and poor outcomes leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No